CLINICAL TRIAL: NCT00744393
Title: The Effect of Sodium Oxybate on Sleep Architecture in Critically Ill Patients: A Double-Blind, Crossover Pilot Study
Brief Title: The Effect of Sodium Oxybate on Sleep Architecture
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor pulled funding secondary to economy issues
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEMC-8479
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Mechanically Ventilated ICU Patients
Keywords: sleep; critically ill; mechanical ventilation
MeSH Terms: conditions — Critical Illness | interventions — Sodium Oxybate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Active drug
  Interventions: Drug: sodium oxybate
- P (Placebo Comparator): Placebo drug
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: sodium oxybate — The dose of sodium oxybate will be 4.5g every 4 hours x 2 doses. The first dose of study medication will be given at 10pm followed by the next dose four hours later and crossed over the next day
  Other Names: XYREM
  Arms: A
Drug: placebo — The dose of placebo sodium oxybate will be 4.5g every 4 hours x 2 doses. The first dose of study medication will be given at 10pm followed by the next dose four hours later and then crossed over the next day
  Other Names: Xyrem
  Arms: P

SUMMARY:
The purpose of this study is to determine what effect sodium oxybate has on the functions of sleep in mechanically ventilated, critically ill patients hospitalized in an intensive care unit.

DETAILED DESCRIPTION:
Sleep is disrupted in the critically ill and may lead to impaired neurocognitive function, decreased immune function, increased protein catabolism, and may compromise the ability to wean patients from mechanical ventilation. Critically ill patients may appear to sleep throughout most of their stay, but their quality of sleep is different from that of a normal healthy subject.Critically ill patients spend more time in the wakefulness stages of sleep (Stage 1 and 2) at the expense of the restorative stages (Stage 3 and 4) and REM sleep. These patients also experience an increased number of arousals and awakenings. Various factors are thought to be the cause of abnormal sleep architecture: ICU environment, pain, illness severity, psychosocial stress, medications, and mechanical ventilation.

Sodium oxybate (Xyrem®) is the sodium salt of the central nervous system depressant γ-hydroxybutyric acid (GHB) and is currently approved for use in narcoleptic patients to improve cataplexy and excessive daytime sleepiness.

Studies evaluating the use of sodium oxybate in narcoleptic patients suggest that sodium oxybate is effective at increasing slow-wave sleep, sleep efficiency, sleep latency, and REM-sleep efficiency, while also decreasing REM-sleep latency, stage 1 NREM sleep and sleep fragmentation.3, 16-19 Currently there is a lack of data evaluating the effects of sodium oxybate on sleep in critically ill patients. Obtaining evidence that sodium oxybate improves sleep architecture in the critically ill, may provide the foundation to complete future studies evaluating the effect of sodium oxybate on clinical outcomes such as duration of mechanical ventilation and length of ICU stay. Based on sodium oxybate's ability to improve sleep architecture in narcoleptic patients along with the fact that critically ill patients have similar disrupted sleep architecture, it's postulated that sodium oxybate may improve the sleep architecture in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Mechanically ventilated ≥ 24º on an AC mode
* Placement of enteral or gastric tube (Note: these tubes will not be placed exclusively for the purposes of the study.)
* Tolerating enteral nutrition via either the stomach or small intestine (≥20mL/hr for ≥ 12 hours)

Exclusion Criteria:

* Anticipated duration of mechanical ventilation ≤72º (as per MICU team estimate)
* Riker SAS ≤ 2 (as determined by patient's nurse and/or study investigator)
* History of irreversible brain disease consistent with severe dementia based on MICU service admission note
* Admitted with a primary neurological condition (e.g. intracranial hemorrhage)
* History of seizure disorder or intracranial surgery
* History of myocardial infarction in prior 6 months
* Pregnancy (all women of child bearing potential will undergo a serum pregnancy test prior to study consent)
* Administration of a scheduled benzodiazepine as either a continuous drip or given by IVP
* Acute alcohol withdrawal
* AST/ALT >2 times ULN, INR >2 or T bilirubin > 1.5
* Current or prior use of sodium oxybate in the -past 30 days.
* Hypernatremia with a serum sodium >150
* Current use of the following hypnotics: barbiturates, melatonin, zolpidem, eszopiclone, or zaleplon
* Use of neuromuscular blocking agents
* Allergy to sodium oxybate
* Known succinic semialdehyde dehydrogenase deficiency
* History of periodic limb movement disorder.
* A prognosis considered to be hopeless (as per MICU team)
* Inability to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
To gain a better understanding of the effect of sodium oxybate on the following components of sleep architecture: % time in sleep stage and arousals and awakenings | 72 hours

SECONDARY OUTCOMES:
To observe any short-term adverse effects of sodium oxybate in mechanically ventilated ICU patients | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn D'Ambrosio, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States